CLINICAL TRIAL: NCT00578604
Title: Non-Invasive Assessment of Wound Healing With Optical Methods
Status: Completed | Type: Observational
Sponsor: Drexel University College of Medicine (Other)
Responsible Party: Sponsor
Organization: Drexel University (Other)
Other Study IDs: 17035
Record Dates: First submitted 2007-12-20; First posted 2007-12-21 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Diabetic Foot Ulcers
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with a diabetic wound: Patients with a diabetic wound
  Interventions: Device: diffuse near infrared spectroscopy measurements
- Control: Patients without a diabetic wound
  Interventions: Device: diffuse near infrared spectroscopy measurements

INTERVENTIONS:
Device: diffuse near infrared spectroscopy measurements — Measure blood flow to diabetic wounds

SUMMARY:
The objective of this project is to further the development of a non-invasive optically based NIR (Near Infrared) device to enable the quantitative diagnosis, monitoring and treatment optimization of chronic wounds (especially diabetic) in a clinical setting. The end goal of this project is a portable and compact device that would be simple to operate by minimally trained health care personnel. Our animal studies have shown that the early healing of chronic wounds can be characterized by absorption and scattering of light at near infrared wavelengths ranging from 680 nm to 950 nm. If our project is successful we will be providing the clinician the ability to predict if a wound is healing and if a particular treatment is successful in accelerating healing before any changes are observed by wound size contraction or other visible clinical signs. Our hope is that the fNIR optical device will provide conclusive therapeutic treatment information as early as 5 weeks after initial evaluation, before it would be obvious on gross examination of the patient.

ELIGIBILITY:
Healthy Subject inclusion criteria

* Subjects must be 18-65 years of age
* Subjects must have no history of diabetes
* Subjects must have no history of vascular disease
* Subjects must have no findings of vascular disease on physical examination
* Subjects who are not allergic to Tegaderm

Patient Subject inclusion criteria:

* Subjects must be 18-65 years of age
* Subjects must have documented diabetes mellitus for at least 6 months.
* Subjects must have at least one documented chronic wound for a minimum 8 weeks.
* A chronic wound is defined as any wound that has not healed after 8 weeks and has a minimum surface area of 1cm2. There is no maximum wound size.
* Wound(s) must be secondary to the complications of diabetes, including vascular disease neuropathy, or both.
* Wounds must be on the ankles or feet
* Subjects who are not allergic to Tegaderm

EXCLUSION CRITERIA

* Subject must not be <18 or >65 years of age
* Subjects with major infections, abscesses, or untreated osteomyelitis will be excluded until appropriately treated.
* Subjects will not be excluded based upon the existence of other co-morbidities associated with chronic diabetes, including retinopathy, nephropathy, peripheral neuropathy, or cardiovascular disease except as follows:
* Subjects who have moderate to severe vascular insufficiency (defined as ankle brachial index <0.75 or toe-brachial index <0.5)
* Subjects who are unable to return for weekly follow-up appointments will not be included.
* Pregnant or lactating people will not be invited to participate.
* Subjects who are allergic to Tegaderm

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Recruited patients will be patients with diabetes who have chronic wounds and will likely have other co-morbidities associated with chronic diabetes.
  Control subjects do not have diabetes and do not have wounds.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2007-09; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
diffuse near infrared spectroscopy measurements | 3 years
  The end goal of this project is a portable and compact device that would be simple to operate by minimally trained health care personnel and is comparable to SOC doppler.

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Weingarten, M.D., Principal Investigator — Drexel University College of Medicine
Locations (1):
- Drexel University College of Medicine Wound Care Center, Philadelphia, Pennsylvania, United States